CLINICAL TRIAL: NCT00709358
Title: Health Economic Evaluation of Rapid Detection of Bacteraemia and Fungemia by Real Time PCR for Cases of Febrile Neutropenia, Suspicion of Endocarditis and Severe Sepsis in Intensive Care Units
Brief Title: Diagnosis of Septicaemia by Detection of Microbial DNA in Blood in Severe Infections
Acronym: EVAMICA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P070308
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-05

CONDITIONS: Febrile Neutropenia; Endocarditis; Severe Sepsis
Keywords: bacteria; fungi; real time PCR; adequate antimicrobial therapy; microbial DNA; microbial diagnosis
MeSH Terms: conditions — Febrile Neutropenia; Endocarditis; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Detection by blood culture
  Interventions: Other: detection of microbial DNA in blood by blood culture
- 1 (Experimental): Test LightCycler SeptiFast® (Roche)
  Interventions: Other: Detection of microbial DNA in blood by SeptiFast®

INTERVENTIONS:
Other: Detection of microbial DNA in blood by SeptiFast® — The LightCycler® SeptiFast Test, the innovative real-time PCR test from Roche Diagnostics, is designed to detect and identify the 25 most important bacterial and fungal species causing bloodstream infections within just a few hours. The LightCycler® SeptiFast Test detects the pathogenic bacteria and fungi directly from whole blood without the need for prior incubation or culture steps.
  Rapid detection and identification of bacterial and fungal DNA, directly from a 1.5 ml whole blood sample, without prior incubation or culture steps in less than 6 hours.
  Arms: 1
Other: detection of microbial DNA in blood by blood culture — A blood culture is a test to find an infection in the blood. Most bacteria can be seen in the culture in 2 to 3 days, but some types can take 10 days or longer to show up. Fungus can take up to 30 days to show up in the culture.
  Arms: 2

SUMMARY:
The primary purpose is to improve and quicken the microbial diagnosis in severe infections, since only one third of the cases are documented by blood cultures and adequate anti-infective therapy in the 48 hours reduced mortality and morbidity.

Our hypothesis is that detection of microbial DNA in blood by real time PCR may increase the number of cases diagnosed for bacteraemia or fungemia and shorten the time to positive results, which will provide information for an adequate anti-infectious therapy.

DETAILED DESCRIPTION:
We will evaluate the advantage of adding the molecular test to the microbial investigations usually done (blood cultures and others) in cases of febrile neutropenia, suspicion of infective endocarditis and severe sepsis in intensive care units.

This is a prospective study conducted in 18 sites (7 in the Paris area and 11 all over France) which will enrolled about 2000 patients over 18 years. Sites are randomized for starting with a 6-month period performing the test or 6-month period without the test (control time with the standard of care).

Primary outcome are the number of patients with documented bacteraemia or fungemia. Secondary outcome are (1) the number of patients with an adequate anti-infective therapy and how long it happens after the diagnosis, (2) mortality, (3) new complicated infection, (4) number of investigations (microbial and non microbial) done for the etiological diagnosis, and global hospitalization costs.

The advantage of the new test will be evaluated per protocol and with an intend to treat analyses. We hypothesized that the new test will bring 15% more microbial diagnosis than the standard of care. Consequently, and according to the number of sites interested in the study, 166 to 2500 patients will be enrolled with 480 to 750 patients with febrile neutropenia, 1000 to 1500 patients with severe sepsis in Intensive Care Units (ICU). Patients with suspicion of infective endocarditis will be evaluated for the number of diagnosis of true endocarditis according to Duke Criteria, and the time to diagnosis.

Health economic evaluation will compare the costs of hospitalization, microbial investigations including the new test, other non clinical investigations and consequences on the organization.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Written signed and dated inform consent
* First time with fever observed in a neutropenic patient
* Severe sepsis in a patient hospitalized in ICU
* Suspicion of infective endocarditis
* Microbial investigation from Monday to Friday

Exclusion Criteria:

* Not affiliated to Health Insurance (social security)
* Included in another interventional trial testing microbial DNA detection during the time "without Septifast®"
* Included in another clinical trial for which the clinician assumes that it will not be possible to prescribe an anti-infectious therapy adequately to microbial detection in the blood
* Patient previously included in the protocol
* Sepsis with a microbial diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Number of bacteraemia and of fungemia - overall - each condition | max Day 30

SECONDARY OUTCOMES:
Number of patients with adequate anti-infective therapy | at day 30
Adequate anti-infective therapy | at 24h, 48h, > 48h
Time between sampling for microbial investigation and positive results relevant for the diagnosis | between sampling for microbial investigation and positive results
Mortality | at Day 30
Sepsis chock, secondary infectious focus | at Day 30
For neutropenia cases, number of patients who evaluated with a clinical focus of infection | at day 30
Diagnosis of endocarditis | at Day 45
Number of non clinical investigations (microbial and non microbial) | at day 30
Length of hospital stay | at day 30

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle CAMBAU, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris; René COURCOL, PH, Principal Investigator — CHRU LILLE
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Cambau E, Durand-Zaleski I, Bretagne S, Brun-Buisson C, Cordonnier C, Duval X, Herwegh S, Pottecher J, Courcol R, Bastuji-Garin S; EVAMICA study team. Performance and economic evaluation of the molecular detection of pathogens for patients with severe infections: the EVAMICA open-label, cluster-randomised, interventional crossover trial. Intensive Care Med. 2017 Nov;43(11):1613-1625. doi: 10.1007/s00134-017-4766-4. Epub 2017 Apr 3. PMID 28374097